CLINICAL TRIAL: NCT00636467
Title: Evaluation of the Technique of Axillary Sentinel Lymph Node (SLN) Detection in Breast Cancers > 2 cm
Brief Title: Axillary Sentinel Lymph Node Detection in Breast Cancers > 2 cm
Acronym: GAS2PLUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: PHRC 2007: financial support (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GAS2PLUS; ET2007-045
Record Dates: First submitted 2008-02-08; First posted 2008-03-14 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer (tumors> 2 cm); Detection; Axillary sentinel lymph node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No label (Experimental): Injection of Nanocis® or Nanocoll® (Tc-colloid) on the day before surgery followed by lymphoscintigraphy (long protocol, method n°1) or injection of Nanocis® or Nanocoll® on the morning of the surgery followed by lymphoscintigraphy at least 2h30 later (short protocol, method n° 2)
  Interventions: Other: No name

INTERVENTIONS:
Other: No name — Injection of Nanocis® or Nanocoll® on the day before surgery followed by lymphoscintigraphy (long protocol, method n°1) or injection of Nanocis® or Nanocoll® on the morning of the surgery followed by lymphoscintigraphy at least 2h30 later (short protocol, method n° 2)

SUMMARY:
The purpose of this study is to evaluate the quality criteria of the SLN detection technique in breast cancer patients with a tumor size (clinical measurement) greater than 2 centimeters (rate of false negatives, rate of detection).

Eligible patients will only be registered (no randomization). The estimated inclusion period is approximately 24 months. The duration of the research is 25 months (24 months for patient inclusion + 1 month for reception of results). The maximum participation duration of each patient is 1 month.

The number of patients required in this multicentric and prospective study is 240 (16 participating centers).

DETAILED DESCRIPTION:
Axillary node extension is one of the major prognostic factors in breast cancer. Axillary dissection of Berg level I and II nodes is the validated method to obtain information on lymph node invasion, but it is associated with important morbidity.

Sentinel lymph node assessment (SLN) was developed to select patients likely not to have axillary node extension using a technique less invasive than conventional dissection. Axillary dissection is restricted to patients with undetected or metastatic SLN.

SLN detection involves subareolar or peri-tumoral injection of lymphotropic contrast agents which map the regional lymphatic drainage pattern of the tumor.

This technique allows an optimization of histopathological analysis: the pathologist must analyze only two nodes on average (instead of 10-15), allowing the examination of numerous tissue sections and the development of specific techniques such as immunohistochemistry.

The principal indicators of success for the technique are the detection rate, the false negative rate and the number of SLN sampled.

The assessment of feasibility is based on concomitant histopathological analysis of the SLN and of complementary lymph nodes.

There is no consensus in the literature on the SLN technique to be used for tumors with clinical size superior to 2 cm in diameter.

The aim of this prospective, multicentric study is to evaluate the performance of the SLN technique, in terms of detection rate and false negative rate, for patients with tumors greater than 2 cm (clinical measurement).

A homogeneous technique with "combined", colorimetric and isotopic SLN detection with subareolar or peri-tumoral injection will be used. This consensus "combined" technique has been validated by all investigators. The histopathological procedure will also be homogeneous, and validated within the group of pathologists of the Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC). Breast surgery will either be a mastectomy or conservative treatment.

The primary objective of the study is to evaluate the quality criteria of the SLN detection technique in breast cancer patients with a tumor size (clinical measurement) greater than 2 centimeters (rate of false negatives, rate of detection).

The secondary objectives are:

* Evaluation of the number of SLN sampled per patient,
* Lymphoscintigraphic evaluation of the pattern of lymphatic drainage in breast tumors > 2 centimeters,
* Precise histopathological description of the SLN sampled and of axillary nodes of levels I and II.

Evaluation criteria:

The primary criterion is the rate of false negatives, determined by the ratio of the number of patients with detected but negative SLN to the total number of positive non-sentinel nodes at the time of axillary dissection of levels I and II (patients classified as N+ according to the TNM system).

This rate will be determined after calculation of the detection rate, determined by the ratio of the number of patients evaluated on the total number of patients.

In agreement with international recommendations, the expected rate of false negatives should be < 5 % with a detection rate > 85 %.

Secondary criteria include:

* Total number of sampled SLN per patient,
* Lymphoscintigraphy: detection of SLN by means of extra-axillary markings,
* Histopathological results:

  * SLN: metastases, capsular breach, micro metastases, isolated cells,
  * Dissection: number of positive nodes.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years
* Patient with invasive unifocal breast cancer with tumor size > 2 cm at initial examination (clinical examination and/or imaging)
* Preoperative histological diagnosis of infiltrating mammary carcinoma
* No lymph node at clinical examination
* No treatment for this cancer before surgery
* Mandatory affiliation with a social security system
* Written, signed informed consent

Exclusion Criteria:

* No invasive breast cancer
* Breast tumor =< 2 cm
* Preoperative histological diagnosis other than infiltrating mammary carcinoma
* Multifocal breast cancer
* Inflammatory breast cancer
* Metastatic cancer
* History of homolateral breast surgery
* History of allergic disorders
* History of homolateral breast cancer
* Difficult follow-up
* Pregnant or lactating woman
* Previous inclusion in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Quality criteria of the SLN detection technique | 1 month

SECONDARY OUTCOMES:
Total number of sampled SLN per patient | 1 month
Detection of SLN by means of extra-axillary markings (lymphoscintigraphy) | 1 month
Histopathological results (SLN) | 1 month
Histopathological results (dissection) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hervé MIGNOTTE, MD, Principal Investigator — Centre Leon Berard, Lyon
Locations (22):
- France (22):
  - Centre Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - CH Boulogne sur Mer, Boulogne-sur-Mer
  - CH Calais, Calais
  - Clinique des 2 Caps, Coquelles
  - Clinique des Acacias, Cucq
  - Clinique Pasteur, Guilherand-Granges
  - Centre Oscar Lambret, Lille
  - Hôtel Dieu, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CH Arrondissement Montreuil sur Mer, Rang-du-Fliers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - CHRU Saint Etienne, Saint-Etienne
  - Centre René Gauducheau, Saint-Herblain
  - CMCO, Saint-Martin-Boulogne
  - Institut Claudius Régaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Bonadonna G, Valagussa P, Moliterni A, Zambetti M, Brambilla C. Adjuvant cyclophosphamide, methotrexate, and fluorouracil in node-positive breast cancer: the results of 20 years of follow-up. N Engl J Med. 1995 Apr 6;332(14):901-6. doi: 10.1056/NEJM199504063321401. PMID 7877646
- [Background] Ivens D, Hoe AL, Podd TJ, Hamilton CR, Taylor I, Royle GT. Assessment of morbidity from complete axillary dissection. Br J Cancer. 1992 Jul;66(1):136-8. doi: 10.1038/bjc.1992.230. PMID 1637663
- [Background] Ververs JM, Roumen RM, Vingerhoets AJ, Vreugdenhil G, Coebergh JW, Crommelin MA, Luiten EJ, Repelaer van Driel OJ, Schijven M, Wissing JC, Voogd AC. Risk, severity and predictors of physical and psychological morbidity after axillary lymph node dissection for breast cancer. Eur J Cancer. 2001 May;37(8):991-9. doi: 10.1016/s0959-8049(01)00067-3. PMID 11334724
- [Background] Kissin MW, Querci della Rovere G, Easton D, Westbury G. Risk of lymphoedema following the treatment of breast cancer. Br J Surg. 1986 Jul;73(7):580-4. doi: 10.1002/bjs.1800730723. PMID 3730795
- [Background] Giuliano AE, Kirgan DM, Guenther JM, Morton DL. Lymphatic mapping and sentinel lymphadenectomy for breast cancer. Ann Surg. 1994 Sep;220(3):391-8; discussion 398-401. doi: 10.1097/00000658-199409000-00015. PMID 8092905
- [Background] Krag DN, Weaver DL, Alex JC, Fairbank JT. Surgical resection and radiolocalization of the sentinel lymph node in breast cancer using a gamma probe. Surg Oncol. 1993 Dec;2(6):335-9; discussion 340. doi: 10.1016/0960-7404(93)90064-6. PMID 8130940
- [Background] Glass EC, Essner R, Giuliano AE. Sentinel node localization in breast cancer. Semin Nucl Med. 1999 Jan;29(1):57-68. doi: 10.1016/s0001-2998(99)80030-0. PMID 9990684
- [Background] Turner RR, Ollila DW, Krasne DL, Giuliano AE. Histopathologic validation of the sentinel lymph node hypothesis for breast carcinoma. Ann Surg. 1997 Sep;226(3):271-6; discussion 276-8. doi: 10.1097/00000658-199709000-00006. PMID 9339933
- [Background] McMasters KM, Tuttle TM, Carlson DJ, Brown CM, Noyes RD, Glaser RL, Vennekotter DJ, Turk PS, Tate PS, Sardi A, Cerrito PB, Edwards MJ. Sentinel lymph node biopsy for breast cancer: a suitable alternative to routine axillary dissection in multi-institutional practice when optimal technique is used. J Clin Oncol. 2000 Jul;18(13):2560-6. doi: 10.1200/JCO.2000.18.13.2560. PMID 10893287
- [Background] Weaver DL, Krag DN, Ashikaga T, Harlow SP, O'Connell M. Pathologic analysis of sentinel and nonsentinel lymph nodes in breast carcinoma: a multicenter study. Cancer. 2000 Mar 1;88(5):1099-107. PMID 10699901
- [Background] Tafra L, McMasters KM, Whitworth P, Edwards MJ. Credentialing issues with sentinel lymph node staging for breast cancer. Am J Surg. 2000 Oct;180(4):268-73. doi: 10.1016/s0002-9610(00)00466-9. PMID 11113433
- [Background] McMasters KM, Wong SL, Chao C, Woo C, Tuttle TM, Noyes RD, Carlson DJ, Laidley AL, McGlothin TQ, Ley PB, Brown CM, Glaser RL, Pennington RE, Turk PS, Simpson D, Edwards MJ; University of Louisville Breast Cancer Study Group. Defining the optimal surgeon experience for breast cancer sentinel lymph node biopsy: a model for implementation of new surgical techniques. Ann Surg. 2001 Sep;234(3):292-9; discussion 299-300. doi: 10.1097/00000658-200109000-00003. PMID 11524582
- [Background] Orr RK, Hoehn JL, Col NF. The learning curve for sentinel node biopsy in breast cancer: practical considerations. Arch Surg. 1999 Jul;134(7):764-7. doi: 10.1001/archsurg.134.7.764. PMID 10401830
- [Background] Bedrosian I, Reynolds C, Mick R, Callans LS, Grant CS, Donohue JH, Farley DR, Heller R, Conant E, Orel SG, Lawton T, Fraker DL, Czerniecki BJ. Accuracy of sentinel lymph node biopsy in patients with large primary breast tumors. Cancer. 2000 Jun 1;88(11):2540-5. doi: 10.1002/1097-0142(20000601)88:113.0.co;2-a. PMID 10861431
- [Background] Chung MH, Ye W, Giuliano AE. Role for sentinel lymph node dissection in the management of large (> or = 5 cm) invasive breast cancer. Ann Surg Oncol. 2001 Oct;8(9):688-92. doi: 10.1007/s10434-001-0688-y. PMID 11597008
- [Background] Lelievre L, Houvenaeghel G, Buttarelli M, Brenot-Rossi I, Huiart L, Tallet A, Tarpin C, Jacquemier J. Value of the sentinel lymph node procedure in patients with large size breast cancer. Ann Surg Oncol. 2007 Feb;14(2):621-6. doi: 10.1245/s10434-006-9232-4. Epub 2006 Nov 12. PMID 17103062
- [Background] Schwartz GF, Giuliano AE, Veronesi U; Consensus Conference Committee. Proceedings of the consensus conference on the role of sentinel lymph node biopsy in carcinoma of the breast, April 19-22, 2001, Philadelphia, Pennsylvania. Cancer. 2002 May 15;94(10):2542-51. doi: 10.1002/cncr.10539. No abstract available. PMID 12173319
- [Background] Lyman GH, Giuliano AE, Somerfield MR, Benson AB 3rd, Bodurka DC, Burstein HJ, Cochran AJ, Cody HS 3rd, Edge SB, Galper S, Hayman JA, Kim TY, Perkins CL, Podoloff DA, Sivasubramaniam VH, Turner RR, Wahl R, Weaver DL, Wolff AC, Winer EP; American Society of Clinical Oncology. American Society of Clinical Oncology guideline recommendations for sentinel lymph node biopsy in early-stage breast cancer. J Clin Oncol. 2005 Oct 20;23(30):7703-20. doi: 10.1200/JCO.2005.08.001. Epub 2005 Sep 12. PMID 16157938
- [Result] Edwards M, Giuliano A, Reintgen D, Tafra L. Consensus statement on guidelines for performance of sentinel lymph node biopsy for breast cancer. Am Soc Breast Surg Q. Press Release, 1998 ;Fall :3